CLINICAL TRIAL: NCT04078308
Title: Phase I/II Clinical Trial to Examine the Safety and Efficacy of Transplantation of Mesenchymal Stem Cells in New-onset Type 1 Diabetes Patients
Brief Title: Mesenchymal Stem Cells Transplantation in Newly Diagnosed Type-1 Diabetes Patients
Acronym: MSCTXT1DM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other); Iranian Stem Cell Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RI-SCBT-94000019; IRCT2016070428786N1 (Registry Identifier: Iranian Registry of Clinical Trials (IRCT)); 94000019 (Other Grant/Funding Number: Royan Institute); REP-441 (Other Grant/Funding Number: Iranian Stem Cell Council, Vice-presidency for Science and Technology, Presidency of the Islamic Republic of Iran)
Record Dates: First submitted 2019-06-24; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; Cell Transplantation; Autologous Transplantation; Mesenchymal Stem Cell
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells Transplantation (Experimental): The patients with Type 1 Diabetes, who will receive Intravenous injection of autologous bone-marrow derived mesenchymal stem cells
  Interventions: Biological: Intravenous Injection of autologous mesenchymal stem cells
- Placebo (Placebo Comparator): The patients with Type 1 Diabetes, who will receive intravenous injection of normal saline (sodium chloride 0.9%)
  Interventions: Other: Intravenous injection of placebo

INTERVENTIONS:
Biological: Intravenous Injection of autologous mesenchymal stem cells — Intravenous injection 1 millions of bone-marrow derived autologous Mesenchymal Stem Cells (MSCs) per kg of patient's body weight in each dose, weeks 0 & 3
  Arms: Mesenchymal Stem Cells Transplantation
Other: Intravenous injection of placebo — Intravenous injection of normal saline (sodium chloride 0.9%)
  Arms: Placebo

SUMMARY:
Study Objects: Diabetes is an autoimmune disease which is mainly caused an immune reaction to beta cells in the pancreas. In this study, mesenchymal stem cells will be used for immune response modulation and improving regeneration. Study design and method: In a Triple blinded randomized placebo-controlled phase I/II clinical trial, 20 patients with newly diagnosed type-1 diabetes who would be visited in Children's Growth and Development Research Center of Tehran University of Medical Sciences and Royan Institute Cell Therapy Center, would be assessed through two groups including the case group and the placebo group. Participants: Patients of both sexes in a range of 8 to 40 years old who have been diagnosed to have type-1 diabetes in no more than 6 weeks, antibody against beta cells diagnosed in their blood, fasting c-peptide more than or equal to 0.3 ng/ml, and are not suffered from other acute or chronic diseases and cancers, would be studied. Interventions: Intravascular transplantation of autologous mesenchymal stem cells in the case group; placebo injection in the control group. Outcome variables: safety and efficacy.

DETAILED DESCRIPTION:
Diabetes is an autoimmune disease which is mainly caused by an immune reaction to beta cells in the pancreas. Today, insulin injection is a routine treatment for diabetes. Although injected insulin maintains blood glucose, this method cannot result in physiologic reaction to blood glucose changes. Moreover, patients are encountered with diabetes complications like neuropathy, nephropathy, visual and cardiovascular problems, and hypoglycemic unawareness. Therefore, based on previous studies, a treatment option that leads to pancreatic beta cell restoration and inhibits the immune response to these cells could be a hopeful clinical choice. In this clinical trial, autologous bone marrow-derived mesenchymal stem cells will be used for immune response modulation and improving regeneration. Hence, based on inclusion and exclusion criteria, 20 patients with type-1 diabetes will be selected and after clarifying the procedure and fulfilling the agreement to participate in this trial, they will be sorted in two groups. Bone marrow is aspirated from patients bone and after isolation of Mesenchymal stem cells and characterization of these cells, patients in case group will be intravenously injected by 1 million autologous mesenchymal stem cells per kg of patient's body weight in each dose in week 0 and 3, whereas the control group receives a placebo. Then patients will be followed up for 1 year. During this time, different parameters would be evaluated in weeks 1, 2,4, and Months 2,3,6,9 and 12. Laboratory screenings will be done during this period to evaluate the safety and efficacy of this treatment.

ELIGIBILITY:
Inclusion criteria:

* Type 1 diabetes detection in less than 6 weeks
* Diabetes diagnosis according to American Diabetes Association (ADA)
* Presence of Antibodies against pancreatic beta cells
* Fasting C-peptide ≥ 0.3 ng/ml

Exclusion Criteria

* Pregnancy or breastfeeding
* Cancer
* Any acute or severe disease (According to physicians' diagnosis: such as cardiac, pulmonary, hepatic, kidney, mental, … diseases)
* Positive results for: Human Immunodeficiency Virus (HIV), Human T-Lymphotropic Virus (HTLV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Cytomegalovirus (CMV)
* Immune deficient or hyper aesthesia
* History of severe ketoacidosis

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07-06 (Actual); Primary Completion 2019-09-26 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 12 months after the first infusion
  Safety will be assessed by evaluating patients based on CTCAE (v.5) to assess treatment-related adverse events after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells
Change from baseline number of hypoglycemic Unawareness episodes at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Number of hypoglycemic unawareness episodes will be assessed by evaluating patients' blood glucose monitoring sheets

SECONDARY OUTCOMES:
Change from Baseline Fasting Blood Sugar (FBS) at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing Fasting Blood Sugar (FBS) at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells and compare the results with baseline Fasting Blood Sugar (FBS)
Change from Baseline C-peptide at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing serum C-peptide at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells and compare the results with baseline serum C-peptide level
Change from Baseline HbA1C at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing HbA1C at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells and compare the results with baseline HbA1C
Change from Baseline 2-hour postprandial blood glucose at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing 2-hour postprandial blood glucose at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells and compare the results with baseline 2-hour postprandial blood glucose
Change from Baseline daily dose of exogenous insulin injected by patients (IU/kg/day) at 12 Months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Exogenous Insulin requirement of patients will be measured based on their daily insulin injection report sheets, total injected insulin units per day will be divided by patient's weight in order to be comparable between different patients.
Change from baseline Lability Index (LI) at 12 Months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing 2 weeks of blood glucose report sheets, calculation is based on the changes in blood glucose levels over time
Change from Baseline SF-36 Quality of life (QOL) questionnaire score at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing change in patients' Quality of life by answering SF-36 questionnaire before transplantation and 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells; This questionnaire asks about general aspects of patients' life.
  The results would be reported as the total score and the scale range is from 0% to 100%. 0% is considered as worse condition and 100% is considered as the best condition.
Change from Baseline Diabetes Specific Quality of life (DQOL) questionnaire score at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing change in patients' Quality of life by answering Diabetes Specific Quality of Life (DQOL) questionnaire before transplantation and 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells; This questionnaire asks about different aspects of patients' life in relation to diabetes.
  The results would be reported as the total score and the scale range is from 0% to 100%. 0% is considered as worse condition and 100% is considered as the best condition.
Changes from baseline Autoantibodies levels in patients' blood at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing patients Islet Cell Antibodies (ICA), Glutamic Acid Decarboxylase Antibodies (GADA), Insulinoma-Associated protein-2 Antibodies (IA-2A) levels after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells
Changes from baseline serum cytokines levels in patients' blood at 12 months after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells | 12 months after the first infusion
  Assessing serum cytokines levels of patients after intravenous transplantation of autologous bone marrow derived Mesenchymal Stem Cells

CONTACTS AND LOCATIONS:
Overall Officials: Abdolhossein Shahverdi, PhD, Study Chair — Royan Institute, ACECR, Tehran, I.R. Iran; Hossein Baharvand, PhD, Study Director — Department of Stem Cells Biology and Technology, Cell Science Research Center, Royan Institute for Stem Cells Biology & Technology, ACECR, Tehran, I.R. Iran; Ali Rabbani, MD, Study Director — Tehran University of Medical Sciences, Tehran, I.R. Iran; Ensiyeh Hajizadeh saffar, MD,PhD, Principal Investigator — Department of Stem Cells Biology and Technology, Cell Science Research Center, Royan Institute for Stem Cells Biology & Technology, ACECR, Tehran, I.R. Iran
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Izadi M, Sadr Hashemi Nejad A, Moazenchi M, Masoumi S, Rabbani A, Kompani F, Hedayati Asl AA, Abbasi Kakroodi F, Jaroughi N, Mohseni Meybodi MA, Setoodeh A, Abbasi F, Hosseini SE, Moeini Nia F, Salman Yazdi R, Navabi R, Hajizadeh-Saffar E, Baharvand H. Mesenchymal stem cell transplantation in newly diagnosed type-1 diabetes patients: a phase I/II randomized placebo-controlled clinical trial. Stem Cell Res Ther. 2022 Jun 20;13(1):264. doi: 10.1186/s13287-022-02941-w. PMID 35725652
- See also: Royan Institute webpage — http://www.royaninstitute.org/cmsen/index.php